CLINICAL TRIAL: NCT04797832
Title: Randomized Bilnded Controlled Trial Comparing The Effect of IV Sodium Ferric Gluconate Complex (FERRLECIT R) on Outcome of Patients Undergoing Transcatheter Aortic Valve Implantation (TAVI)
Brief Title: IV Sodium Ferric Gluconate Complex in Patients Undergoing TAVI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Erez Marcusohn MD, Dr, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0438-20 RMB
Record Dates: First submitted 2021-03-09; First posted 2021-03-15 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Iron Deficiency Anemia Due to Blood Loss; Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — ferric gluconate

STUDY DESIGN:
Intervention Model Description: Single blinded randomized control trial.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor is blinded to whether the patient received IV Iron.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator): 100 patients receiving IV Iron during index hospitalisation.
  Interventions: Drug: IV Sodium Ferric Gluconate Complex
- No treatment (No Intervention): 100 patients not receiving IV Iron above standout treatment.

INTERVENTIONS:
Drug: IV Sodium Ferric Gluconate Complex — 125 mg of IV Iron per day to 3 to 5 days according to hospitalisation length.
  Other Names: IV Ferrlecit
  Arms: Treatment

SUMMARY:
Iron deficiency is common among patients undergoing TAVI. It is estimated at 54-79%. Previous non-randomized small trial have shown symptomatic benefit in treating iron deficiency in this group of patients.

The investigators predict, that as IV iron will improve symptoms, quality of life and exercise tolerance in this group of patients.

DETAILED DESCRIPTION:
Iron deficiency (ID) among patients undergoing transcatheter aortic valve implantation (TAVI) is common (54%-79% .These patients suffer from higher mortality, unplanned readmission for worsening heart failure or red blood cell transfusions during the first year after TAVI.IV Iron therapy was found to be feasible in the 56 patients who were treated and showed improvement in symptoms at 30 days follow-up.Anemia in TAVI patients is multifactorial, related to advanced age, frailty, coagulopathy, medications, kidney disease, bleeding, inflammation and ID. The most treatable part is ID.

Iron deficiency (ID) is a common comorbidity in other diseases. In heart failure (HF) patients, it is associated with poor outcome, worsening of New York Heart Association (NYHA) Class, and re-hospitalizations. While the mechanisms and pathophysiology of ID in HF is not well understood, it is presumed to be a combination of impaired absorption, renal dysfunction, hemodilution and drugs that are used for the treatment of HF.

The advantages of (intra-venous) IV ferric carboxymaltose to patients with reduced ejection fraction (HFrEF) with stable chronic heart failure and functional ID has been shown to reduce the risk of hospitalizations up to 60%, improve symptoms, exercise tolerance, functional capacity and overall QoL]. Accordingly, the latest 2016 ESC Guidelines recommended the treatment in patients with HfrEF with reduced ejection fraction (HFrEF) and ID (Class IIA,LOC A). No guidelines recommend IV iron supplementation in TAVI patients.

The two major, placebo-controlled studies, mentioned above (CONFIRM-AF and FAIR-AF) have demonstrated the positive outcomes after correction of ID in stable HF patients, with a well-tolerated IV substance. Furthermore, the effect of treating iron deficiency on quality of life and functional status has already been studied and found useful with various types of intravenous iron in the chronic kidney disease and inflammatory bowel disease.The effect of treating with oral iron supplements has been studied in HF patients with no difference in exercise capacity, symptoms, NT pro BNP, iron stores, Hemoglobin levels or V02 compared to placebo.

In this study the investigators aim to examine the effect of IV iron (ferric gluconate) which is a more affordable IV Iron on patients with ID admitted for TAVI. No randomized trial has been published in this topic to this day.

ELIGIBILITY:
* Inclusion criteria: (All criteria need to be met)

  1. Patients admitted for TAVI.
  2. Hb level 8-14 mg/dl on admission.
  3. No evidence of active bleeding.
  4. Patient provided informed consent.
  5. The patient is able to walk without support for 6 minutes.
  6. LVEF >= 45%
* Exclusion criteria:

  1. Previous allergy or anaphylaxis due to IV Iron.
  2. Active malignancy undergoing treatment.
  3. Status post major surgery involving substantial blood loss in the past 3 months.
  4. Infection indicating IV antibiotics, not including prophylaxis for TAVI.
  5. History of acquired iron overload; known haemochromatosis or first relatives with hemochromatosis; and allergic disorders (asthma, eczema, and anaphylactic reactions).
  6. Hemolytic anemia.
  7. History of chronic liver disease and/or alanine transaminase (ALT) or aspartate transaminase (AST) >3 times the upper limit of the normal range; chronic lung disease; myelodysplastic disorder; and known HIV/AIDS disease.
  8. Recipient of immunosuppressive therapy or renal dialysis. History of erythropoietin, IV iron therapy, and blood transfusion in previous 30 days.
  9. Musculoskeletal limitation that, in the judgement of the investigator, would impair 6-minute walk.
  10. Pregnant or breastfeeding.
  11. Inability to comprehend study protocol.
  12. Parallel participation in another clinical trial.
  13. During TAVI or the day following the procedure:

I. Major complication of death. II. Cardiogenic shock or any other condition requiring IV vasopressors. III. Major bleeding according to BARC 2 criteria or above. IV. Need for more than 2 pack cells during or after the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-10-18 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
6-minute walk change at 1 month. | 30 days.
  6-minute walk change (meters) between baseline and 1 month follow-up.
6-minute walk change at one year. | One year.
  6-minute walk change (meters) between baseline and 1 year follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Erez Marcusohn, MD, Principal Investigator — Cardiology Department, Rambam Health Care Campus,Haifa,Israel
Locations (1):
- Rambam Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No